CLINICAL TRIAL: NCT00336947
Title: Controlled Randomized Trial to Evaluate Efficacy of Adjuvant Chemotherapy Between S-1 and UFT for Locally Advanced Squamous Cell Carcinoma of the Head and Neck: Phase III Study
Brief Title: S-1 or Tegafur-Uracil in Treating Patients With Previously Treated Stage III or Stage IV Head and Neck Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yokohama City University (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: YCU-BRI-HN-05-01; CDR0000486874 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2006-06-13; First posted 2006-06-15 (Estimated); Last update posted 2013-05-15 (Estimated); Status verified 2008-12

CONDITIONS: Head and Neck Cancer
Keywords: stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — Tegafur; Chemotherapy, Adjuvant

INTERVENTIONS:
Drug: tegafur-gimeracil-oteracil potassium
Drug: tegafur-uracil
Procedure: adjuvant therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as S-1 and tegafur-uracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving S-1 or tegafur-uracil after surgery, chemotherapy, biological therapy, and/or radiation therapy may kill any remaining tumor cells. It is not yet known whether S-1 is more effective than tegafur-uracil in treating head and neck cancer.

PURPOSE: This randomized phase III trial is studying S-1 to see how well it works compared with tegafur-uracil in treating patients with previously treated stage III or stage IV head and neck cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the disease-free survival rate in patients with definitively treated stage III or IV squamous cell carcinoma of the head and neck treated with adjuvant chemotherapy comprising S-1 vs tegafur-uracil (UFT).

OUTLINE: This is a randomized, controlled, multicenter study. Patients are stratified according to primary site, disease stage, type of prior definitive treatment, and participating center. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral S-1 once daily on days 1-14. Courses repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity.
* Arm II:Patients receive oral tegafur-uracil (UFT) once daily on days 1-21. Courses repeat every 21 days for 1 year in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 500 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed squamous cell carcinoma of the head and neck (SCCHN)

  * Stage III or IV disease
  * Primary tumor in the mesopharynx, hypopharynx, larynx (except T3 N0 tumors of the glottis), oral cavity, or maxillary sinus
* Completed definitive treatment for SCCHN within the past 3 months, that included any of the following:

  * Surgery
  * Chemotherapy
  * Biologic therapy
  * Radiotherapy (e.g., radiotherapy in combination with chemotherapy or pre- or postoperative radiotherapy)
  * Any other treatment
* No clinical evidence of locoregional tumors or distant metastasis within 3 months after the completion of definitive treatment

PATIENT CHARACTERISTICS:

* ECOG performance status 0-1
* WBC ≥ 3,500/mm^3 AND ≤ 12,000/mm^3
* Neutrophil count ≥ 2,000/mm^3
* Platelet count ≥ 100,000/mm^3
* Hemoglobin ≥ 9 g/dL
* AST and ALT < 100 IU/L
* Bilirubin < 1.5 mg/dL
* Creatinine < 1.2 mg/dL
* No uncontrolled cardiovascular disease
* No interstitial pneumonia or pulmonary fibrosis
* Must have sufficient oral intake

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* No concurrent biologic therapy, radiotherapy, other chemotherapy, or any other therapy

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2006-04; Primary Completion 2012-03 (Estimated)

PRIMARY OUTCOMES:
Disease-free survival

SECONDARY OUTCOMES:
Relapse-free survival
Overall survival
Adverse effects

CONTACTS AND LOCATIONS:
Overall Officials: Mamoru Tsukuda, MD, Study Chair — Yokohama City University
Locations (48):
- Japan (48):
  - Aichi Cancer Center, Nagoya, Aichi-ken
  - Fujita Health University, Toyoake, Aichi-ken
  - Akita University Hospital, Akita, Akita
  - Tokyo Dental College Ichikawa General Hospital, Ichikawa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - University of Fukui Hospital, Fukui-shi, Fukui
  - National Kyushu Cancer Center, Fukuoka, Fukuoka
  - Fukushima Medical University Hospital, Fukushima, Fukushima
  - Gifu University Graduate School of Medicine, Gifu, Gifu
  - Gunma University Graduate School of Medicine, Maebashi, Gunma
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Hyogo Cancer Center, Akashi, Hyōgo
  - National Hospital Organization - Himeji Medical Center, Himeji-shi, Hyōgo
  - Kanazawa Medical University, Kanazawa, Ishikawa-ken
  - Iwate Medical University Hospital, Morioka, Iwate
  - Kagoshima University, Kagoshima, Kagoshima-ken
  - Kagoshima City Hospital, Kagoshima, Kagoshima-ken
  - Yokohama Rosai Hospital, Yokohama, Kanagawa
  - Yokohama City University, Yokohama, Kanagawa
  - Kumamoto University Medical School, Kumamoto, Kumamoto
  - Mie University Graduate School of Medicine, Tsu, Mie-ken
  - Tohoku University Graduate School of Medicine, Sendai, Miyagi
  - Miyazaki Medical College University of Miyazaki, Miyazaki-gun, Miyazaki
  - Tenri Hospital, Tenri, Nara
  - Niigata Prefectural Central Hospital, Jōetsu, Niigata
  - Kawasaki Medical School, Kurashiki, Okayama-ken
  - Osaka General Medical Center, Osaka, Osaka
  - Osaka City University, Osaka, Osaka
  - Kinki University School of Medicine, Sayama, Osaka
  - Saitama Cancer Center, Saitama, Saitama
  - Shimane University Hospital, Izumo, Shimane
  - Seirei Hamamatsu General Hospital, Hamamatsu, Shizuoka
  - Hamamatsu University School of Medicine, Hamamatsu, Shizuoka
  - Saiseikai Utsunomiya Hospital, Utsunomiya, Tochigi
  - Tokyo Medical University Hachioji Medical Center, Hachiōji, Tokyo
  - National Tokyo Medical Center, Menguro-ku, Tokyo
  - Kyorin University School of Medicine - Mitaka Campus, Mitaka-shi, Tokyo
  - Ome Municipal General Hospital, Ome-shi, Tokyo
  - Juntendo University School of Medicine, Tokyo, Tokyo
  - Tokyo Medical and Dental University, Tokyo, Tokyo
  - Nippon Medical School, Tokyo, Tokyo
  - Cancer Institute Hospital of Japanese Foundation for Cancer Research, Tokyo, Tokyo
  - Tokyo Medical University, Tokyo, Tokyo
  - Keio University School of Medicine, Tokyo, Tokyo
  - International Medical Center of Japan, Tokyo, Tokyo
  - Tottori University Hospital, Yonago-shi, Tottori
  - Wakayama Medical University, Wakayama, Wakayama
  - Interdiciplinary Graduate School of Medicine and Engineering, Yamanashi, Yamagata

REFERENCES:
- [Derived] Tsukahara K, Kubota A, Hasegawa Y, Takemura H, Terada T, Taguchi T, Nagahara K, Nakatani H, Yoshino K, Higaki Y, Iwae S, Beppu T, Hanamure Y, Tomita K, Kohno N, Kawabata K, Fukushima M, Teramukai S, Fujii M; ACTS-HNC group. Randomized phase III trial of adjuvant chemotherapy with S-1 after curative treatment in patients with squamous-cell carcinoma of the head and neck (ACTS-HNC). PLoS One. 2015 Feb 11;10(2):e0116965. doi: 10.1371/journal.pone.0116965. eCollection 2015. PMID 25671770